CLINICAL TRIAL: NCT05929248
Title: A Randomized Controlled Trial Aimed at Exploring the Efficacy of Telitacicept in the Treatment of Systemic Lupus Erythematosus Patients With Refractory Thrombocytopenia
Brief Title: Exploring the Therapeutic Effect of Telitacicept on Lupus Erythematosus Complicated With Thrombocytopenia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guanmin Gao (Other)
Responsible Party: Sponsor-Investigator, Guanmin Gao, chief physician, The First Affiliated Hospital of Zhengzhou University
Organization: The First Affiliated Hospital of Zhengzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GGao
Record Dates: First submitted 2023-06-14; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Systemic Lupus Erythematosus
Keywords: lupus erythematosus; Telitacicept; thrombocytopenia
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Thrombocytopenia | interventions — telitacicept

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): conventional treatment plus Telitacicept 160 mg sc per week
  Interventions: Drug: Telitacicept; Drug: conventional therapy
- Control group (Placebo Comparator): Placebo plus conventional treatment
  Interventions: Drug: conventional therapy; Drug: Placebo

INTERVENTIONS:
Drug: Telitacicept — 160mg once a week for 48 weeks
  Other Names: RC18
  Arms: Treatment group
Drug: conventional therapy — Steroid(≤1mg/kg/d) with or without proper immunosuppressants：CTX, MMF, AZA, CsA, FK 506, HCQ, MTX, LEF, SASP etc.
Drug: Placebo — Used once a week in combination with standard treatment
  Arms: Control group

SUMMARY:
The purpose of this study is to evaluate the efficacy of telitacicept in patients with systemic lupus erythematosus and refractory thrombocytopenia

DETAILED DESCRIPTION:
This study is a single center, randomized, controlled trial to evaluate the efficacy of telitacicept in patients with systemic lupus erythematosus complicated with refractory thrombocytopenia.

ELIGIBILITY:
Inclusion Criteria:

1. Meets the 2012 ACR revised standards and meets four or more diagnostic criteria for systemic lupus erythematosus;
2. Refractory thrombocytopenia (defined as receiving at least one course of methylprednisolone pulse therapy or intravenous injection of high-dose immunoglobulin or high-dose glucocorticoid combined with two or more Immunosuppressive drug failed and did not respond to any single drug);
3. SLEENA-SLEDAI score is greater than or equal to 8 points. If anti ds-DNA antibody is positive and/or low complement, SLEENA-SLEDAI score is greater than or equal to 6 points, or PLT count is<10 * 10 ^ 9/L or<30 * 10 ^ 9/L with bleeding tendency;
4. Age greater than or equal to 18 years old and less than or equal to 65 years old;
5. Have a stable SLE treatment plan, and participants should receive standard treatment for at least 30 days before randomization; 6. Positive Antinuclear antibody or anti ds DNA antibody;

7. Sign informed documents.

Exclusion criteria:

Potential subjects who meet the inclusion criteria will be excluded if they meet any of the following criteria:

1. Patients who are allergic to tamoxifen;
2. Patients with severe active infection, history of tuberculosis, malignant tumor, HIV, hepatitis B, hepatitis C, important organs or hematopoietic stem cells/cells/bone marrow transplantation or kidney transplantation;
3. Patients with severe active central nervous system lupus and severe active lupus nephritis
4. Patients with diseases of liver, kidney, heart and other important organs, blood and Endocrine system;
5. Pregnant and lactating women;
6. Have a pregnancy preparation plan in the past year;
7. Those who have merged with other autoimmune diseases;
8. Incomplete case data and missing persons.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
The remission rate of SLE response index at month 12 of treatment | months 12
  Use SRI-4 to represent the response index, with a higher response rate indicating better drug efficacy
Improvement in platelet count | months 12
  Platelet count at month of treatment，Increased platelet count indicates improvement in disease

SECONDARY OUTCOMES:
Percentage of patients with a decrease of ≥ 4 points in the SELENA-SLEDAI score from baseline at months 6 and 12 | months 6 and 12
  A decrease of ≥ 4 points from baseline in the SELENA-SLEDAI score indicates a good drug response effect
Hormone reduction | month 12
  Changes in patient hormone dose from baseline at month 12，reduced hormone dosage indicates improvement in disease
B lymphocyte count | month 12
  Changes in patient B lymphocyte count from baseline at month 12

CONTACTS AND LOCATIONS:
Overall Officials: Gao Guanmin, Principal Investigator — The First Affiliated Hospital of Zhengzhou University